CLINICAL TRIAL: NCT00603954
Title: Allogeneic Hematopoietic Cell Transplantation With HLA-matched Donors : a Phase II Randomized Study Comparing 2 Nonmyeloablative Conditionings
Brief Title: Allogeneic HCT With HLA-matched Donors : a Phase II Randomized Study Comparing 2 Nonmyeloablative Conditionings
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Maastricht University Medical Center (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Yves Beguin, Prof, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJB0702P1
Record Dates: First submitted 2008-01-02; First posted 2008-01-29 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-11

CONDITIONS: Hematological Malignancies
Keywords: Nonmyeloablative conditioning.; Hematological malignancies.; GVHD.
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; Whole-Body Irradiation; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TBI + fludarabine (Active Comparator): Conditioning regimen consisting of fludarabine 30 mg/m2 on days -4, -3 and -2 (total dose 90 mg/m2), followed by a singe dose of 2 Gy TBI administered on day 0, at a low dose-rate (≈ 7 cGy/min), before infusion of cells.
  Interventions: Drug: Conditioning regimen: TBI + Fludarabine
- TLI + ATG (Active Comparator): Conditioning consisting of 8 Gy TLI and ATG. TLI will be administered by linear accelerator at a dose of 80 cGy daily, starting 11 days before transplantation, until a total of 10 doses (800 cGy) has been delivered. The irradiation will consist of a supradiaphragmatic mantle field, a subdiaphragmatic field including an inverted Y and splenic ports, encompassing all major lymphoid organs, including the thymus, spleen, and lymph nodes, as used in the treatment of Hodgkin's disease (Kaplan HS, Cancer Research 26:1268-1276, 1966). The Waldeyer ring is not included. ATG (Thymoglobulin®, Genzyme), at a dose of 1.5 mg/kg/d, will be given intravenously on days -11 through -7.
  Interventions: Drug: Conditioning regimen:TLI (8 Gy) + ATG

INTERVENTIONS:
Drug: Conditioning regimen: TBI + Fludarabine — 2 Gy TBI, Fludarabine 90 mg/m²
  Other Names: total body irradiation (TBI) + fludarabine
  Arms: TBI + fludarabine
Drug: Conditioning regimen:TLI (8 Gy) + ATG — TLI 8 Gy + ATG (Thymoglobulin) 7.5 mg/kg
  Other Names: Total Lymphoid Irradiation (TLI) and Anti-Thymocyte Globulin (ATG)
  Arms: TLI + ATG

SUMMARY:
The present project aims at comparing two nonmyeloablative regimens currently used in 2 major HCT centers in the US for patients with HLA-matched related or unrelated donor: the one from the Seattle group consisting of 2 Gy TBI with fludarabine (90 mg/m²) versus the one from the Stanford group combining 8 Gy TLI with ATG.

DETAILED DESCRIPTION:
I. OBJECTIVES

The present project aims at comparing two nonmyeloablative regimens currently used in 2 major HCT centers in the US for patients with HLA-matched related or unrelated donor: the one from the Seattle group consisting of 2 Gy TBI with fludarabine (90 mg/m²) versus the one from the Stanford group combining 8 Gy TLI with ATG.

II. DESIGN OF THE STUDY

The study is a multicenter, randomized phase II study, comparing two conditioning regimens. Sixty patients with HLA-matched donors will be randomized between the TBI or the DLI regimen. There will be a stratification between centers. There will be a stopping rule for graft rejection > 15% at day 180 (in each group separately), and for nonrelapse mortality > 35% at day 180 (in each group separately). If the stopping rules are not triggered after 60 patients and no statistically significant differences are seen between the 2 arms in terms of acute GVHD, graft rejection and survival, a second cohort of 40 patients will be included.

III. TREATMENT PLAN

III.1. Pre-transplant procedures Peripheral blood mononucleated cells from the patient as well as from the donor will be collected before conditioning, as per standard practice for all routine allogeneic HSC transplants. Part will be cryopreserved in 10 % DMSO and stored at -180°C in liquid nitrogen. The other part will be devoted to identification of specific donor and patient markers to be used in later measurements of chimerism.

III.2. Conditioning regimens The conditioning regimens used will be either the one developed in Seattle (TBI arm) or the one developed by the Stanford group (TLI arm). These 2 regimens have been extensively reported in major medical journals. In the TBI arm, conditioning will consist of fludarabine 30 mg/m2 on days -4, -3 and -2 (total dose 90 mg/m2), followed by a singe dose of 2 Gy TBI administered on day 0, at a low dose-rate (≈ 7 cGy/min), before infusion of cells. In the TLI arm, conditioning will consist of 8 Gy TLI and ATG. TLI will be administered by linear accelerator at a dose of 80 cGy daily, starting 11 days before transplantation, until a total of 10 doses (800 cGy) has been delivered. The irradiation will consist of a supradiaphragmatic mantle field, a subdiaphragmatic field including an inverted Y and splenic ports, encompassing all major lymphoid organs, including the thymus, spleen, and lymph nodes, as used in the treatment of Hodgkin's disease (Kaplan HS, Cancer Research 26:1268-1276, 1966). The Waldeyer ring is not included. ATG (Thymoglobulin®, Genzyme), at a dose of 1.5 mg/kg/d, will be given intravenously on days -11 through -7.

III.3. PBSC collection and transplantation PBSC mobilization and collection in the donor will be performed as per standard practice for all routine allogeneic HSC transplants. This is briefly described below.

The donor will be given SC injections of G-CSF at a dose of 10-15 µg/kg for 6 days (days -5 through 0). Additional doses of G-CSF may be given on days +1 and +2 if the first 2 leukaphereses do not yield sufficient numbers of CD34+ cells. G-CSF will generally be administered :

* In the evening on days -5, -4, -3, -2;
* Before 7:00 on days -1 and 0 (and on days 1 and 2 if necessary). Collection of PBSC will be carried out on day -1 and in the morning on day 0. Leukaphereses will be performed using a continuous flow blood cell separator and following a mononuclear cell collection protocol. The volume of blood processed will be 15-20 liters if donor is an adult or 10 liters/m2 if donor is a child. Anticoagulation will be performed with the ACD-A solution. The PBSC from the first day of harvest will be stored overnight at 4°C in the patient's own plasma. After the second harvest, PBSC from the first and second day of harvest will be infused into the patient.

Based on previous reports suggesting that higher dose of CD34 cells are associated with better outcomes after nonmyeloablative HCT, high doses of CD34+ cells (>6.5 x 106/kg) should be ideally administered. Nevertheless, to limit donor procedures, only two leukaphereses are required. However, in case the required minimal number of cells (3 x 106 CD34+ cells/kg recipient) cannot be obtained with the first two collections, additional leukaphereses should be carried out unless contra-indicated for the donor.

Cells will be infused through a central catheter according to standard procedures.

III.4. Other treatments of the recipient

III.4.1. Immunosuppressive therapy The immunosuppressive regimens used will be the one used in standard practice for routine NM-HCT at our centers, i.e. an association of tacrolimus and mycophenolate mofetil (MMF).

MMF will be administered orally from the evening of day 0 through day 28 (sibling recipients) or day 42 (alternative donor recipients) at the dose of 15 mg/kg t.i.d.

Tacrolimus will be given orally at the dose of 0.06 mg/kg bid starting on day -3. The dose will then be adapted according to through whole blood values following standard procedures (between 15 and 20 ng/ml the first 28 days and between 10-15 ng/ml thereafter). Full doses will be given until day 100 (sibling recipients) or 180 (alternative donor recipients). Doses will then be progressively tapered to be definitely discontinued by day 180 (sibling donors) or 365 (alternative donor recipients) in the absence of GVHD. Tacrolimus may be stopped earlier in case of disease progression or graft rejection or continued longer in case of low donor T-cell chimerism or GVHD.

GVHD will be assessed according to standard criteria. Therapy for acute or chronic GVHD will use standard procedures/current protocols.

III.4.2. Growth factors Growth factors will be used as per standard practice for all routine NM-HCT. No myeloid growth factor will be administered unless the granulocyte count falls below 1000/µl. Patients may then be treated with 5 µg/kg/day of G-CSF to maintain the granulocyte count > 1,000/µl. Erythropoietin may be administered as required.

III.4.3. Infection prophylaxis Infection prophylaxis against bacterial, fungal, viral and parasitic agents will be carried out as per standard practice for all routine NM-HCT.

III.4.4. Donor lymphocyte infusion Donor lymphocyte infusion (DLI) will be given as per standard practice for all routine NM-HCT. DLI may be given in case of poor T-cell chimerism or disease progression according to standard procedures/current protocols.

IV. PATIENTS' FOLLOW-UP

IV.1. Quality controls of cell products

IV.1.1. Peripheral blood of donor on days of PBSC collection As per standard practice for all routine allogeneic PBSC transplants.

IV.1.2. Leukapheresis product As per standard practice for all routine allogeneic PBSC transplants including determination of the number of TNC, CD34, CD3 , CD4 and CD8 cells transplanted.

IV.2. Toxicities of cell infusions Potential toxicities associated with PBSC infusions will be carefully monitored per the standard procedures.

IV.3. Chimerism The chimeric status of hematopoietic cells will be carefully monitored post-transplant, as per standard practice for all routine allogeneic transplants. Donor chimerism will be measured in whole blood as well as bone marrow. In addition, peripheral blood cells will be separated by RosetteSep procedure (Stem Cell Technologies, Vancouver, Canada) to determine the proportion of donor and recipient cells in pure population of T (CD3+) cells. Fluorescent in-situ hybridization (FISH) for X and Y chromosome will be used preferentially for sex-mismatched HCT, while PCR techniques based on short tandem repeat (STR) markers will be used for sex-matched HCT. Pre-transplant donor and recipient peripheral WBC will serve to identify specific markers.

We define complete chimerism as the presence of >95% of T cells of donor origin and mixed chimerism as the presence of 6-94% of T cells of donor origin. Graft rejection is defined as the occurrence of T cell chimerism < 5% and engraftment as the occurrence of more than 5% T cells of donor origin in the first month following the transplant.

The proportion of donor chimerism will be determined at the following time points:

1. peripheral blood :

   * Days 28, 42, 60, 100, 180 and 365 post-transplant : whole blood and CD3+ cells;
   * Analyses on day 60 are only necessary when chimerism is < 80% on days 28 and/or 42;
   * Analyses on whole blood on days 42, 100, 180 and 365 are only necessary when bone marrow analyses are not feasible/successful.
2. bone marrow : • Days 42, 100, 180 and 365 post-transplant : whole bone marrow.

IV.4. Clinical data Patient will be carefully observed and the following clinical parameters will be recorded (see appendices B and C). Appendices B and C should be send not more than 3 months after the patient achieved the target day after HSCT (day 100, day 180, 1-yr, 2-yr, 3-yr, 4-yr and 5-yr) to Frederic Baron at the fax # 32-4-366 8855.

* Incidence, timing and severity of acute GVHD, its treatment and outcome;
* Incidence, timing and severity of chronic GVHD, its treatment and outcome;
* Incidence, timing and severity of cytopenia, its treatment and outcome; number of platelet and RBC transfusions; G-CSF usage;
* Time to achieve 500 neutrophils, 1000 neutrophils, 20 000 platelets and 50 000 platelets;
* Duration of hospitalization, if any;
* Incidence of bacterial infections;
* Incidence of fungal infections;
* Incidence of CMV infections (by quantitative PCR) and CMV disease;
* Incidence of other viral infections;
* Incidence of other infections;
* Evolution of the primary malignant disease : response, relapse, its treatment and outcome;
* Any other serious complication associated with the transplant procedure;
* Death and survival.

IV.5. Immunologic data. In patients transplanted at the university of Liège, immune reconstitution in the patient will be monitored as per standard practice at ULg for all routine allogeneic transplants. For patients transplanted outside of the University of Liège and willing to participate to the immune recovery study, 50 mL of fresh heparinized blood collected on days 42, 100, 180, 365 and 730 can be send at room temperature to Olivier Dengis, Department of Clinical Hematology, CHU Sart-Tilman, B4000 Liège.

ELIGIBILITY:
Inclusion Criteria:

PATIENT

1. Diseases

   Hematological malignancies confirmed histologically and not rapidly progressing:
   * AML in CR (defined as ≤ 5% marrow blasts and absence of blasts in the peripheral blood);
   * MDS with ≤ 5% marrow blasts and absence of blasts in the peripheral blood;
   * CML in CP;
   * MPS not in blast crisis and not with extensive marrow fibrosis,
   * ALL in CR;
   * Multiple myeloma not rapidly progressing;
   * CLL;
   * Non-Hodgkin's lymphoma (aggressive NHL should have chemosensitive disease);
   * Hodgkin's disease with chemosensitive disease.
2. Clinical situations

   * Theoretical indication for a standard allo-transplant, but not feasible because:

     * Age > 50 yrs;
     * Unacceptable end organ performance;
     * Patient's refusal.
   * Indication for a standard auto-transplant: perform mini-allotransplantation 2-6 months after standard autotransplant.
3. Other inclusion criteria

   * Male or female; fertile patients must use a reliable contraception method;
   * Age < 75 yrs;
   * Informed consent given by patient or his/her guardian if of minor age.

DONOR

* Related to the recipient (sibling, parent or child) or unrelated;
* Male or female;
* Any age;
* 10 of 10 (HLA-A, -B, -C, -DRB1, and -DQB1) HLA allele matched;
* Weight > 15 Kg (because of leukapheresis);
* Fulfills criteria for allogeneic PBSC donation according to standard procedures;
* Informed consent given by donor or his/her guardian if of minor age, as per donor center standard procedures.

Exclusion Criteria:

PATIENT

* Any condition not fulfilling inclusion criteria;
* HIV positive;
* Non-hematological malignancy(ies) (except non-melanoma skin cancer) < 3 years before nonmyeloablative HCT.
* Life expectancy severely limited by disease other than malignancy;
* Administration of cytotoxic agent(s) for "cytoreduction" within three weeks prior to initiating the nonmyeloablative transplant conditioning (Exceptions are hydroxyurea and imatinib mesylate);
* CNS involvement with disease refractory to intrathecal chemotherapy.
* Terminal organ failure, except for renal failure (dialysis acceptable)
* Uncontrolled infection;
* Karnofsky Performance Score <70%;
* Patient is a fertile man or woman who is unwilling to use contraceptive techniques during and for 12 months following treatment;
* Patient is a female who is pregnant or breastfeeding;
* Previous radiation therapy precluding the use of 2 Gy TBI or 8 Gy TLI;

DONOR

* Any condition not fulfilling inclusion criteria;
* Unable to undergo leukapheresis because of poor vein access or other reasons.

Max Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Baron, MD, PhD, Study Chair — CHU-ULg; Yves Beguin, MD, PhD, Study Chair — CHU-ULg; Johan Maertens, MD, Principal Investigator — KUL; Koen Theunissen, MD, Principal Investigator — KUL; Harry Schouten, MD, Principal Investigator — Maastricht University Medical Center
Locations (11):
- Belgium (10):
  - AZ Gasthuisberg Leuven, Leuven, Flamish Brabant
  - UZ Gent, Ghent, Flanders Oost
  - University Hospital Mont-Godinne, Godinne, Namur
  - AZ St-Jan, Bruges, West Flanders
  - UZA Stuyvenberg, Antwerp
  - UZA, Antwerp
  - Bordet Institute, Brussels
  - St Luc UCL, Brussels
  - UZ Brussels, Brussels
  - CHU Sart Tilman, Liège
- University Hospital Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Hannon M, Beguin Y, Ehx G, Servais S, Seidel L, Graux C, Maertens J, Kerre T, Daulne C, de Bock M, Fillet M, Ory A, Willems E, Gothot A, Humblet-Baron S, Baron F. Immune Recovery after Allogeneic Hematopoietic Stem Cell Transplantation Following Flu-TBI versus TLI-ATG Conditioning. Clin Cancer Res. 2015 Jul 15;21(14):3131-9. doi: 10.1158/1078-0432.CCR-14-3374. Epub 2015 Mar 16. PMID 25779951
- [Derived] Baron F, Zachee P, Maertens J, Kerre T, Ory A, Seidel L, Graux C, Lewalle P, Van Gelder M, Theunissen K, Willems E, Emonds MP, De Becker A, Beguin Y. Non-myeloablative allogeneic hematopoietic cell transplantation following fludarabine plus 2 Gy TBI or ATG plus 8 Gy TLI: a phase II randomized study from the Belgian Hematological Society. J Hematol Oncol. 2015 Feb 6;8:4. doi: 10.1186/s13045-014-0098-9. PMID 25652604

RESULTS

PARTICIPANT FLOW:
Groups:
- Flu-TBI: Conditioning regimen consisting of fludarabine 30 mg/m2 on days -4, -3 and -2 (total dose 90 mg/m2), followed by a singe dose of 2 Gy TBI administered on day 0, at a low dose-rate (≈ 7 cGy/min), before infusion of cells.
  Conditioning regimen TBI + Fludarabine: 2 Gy TBI, Fludarabine 90 mg/m²
- TLI-ATG: Conditioning consisting of 8 Gy TLI and ATG. TLI will be administered by linear accelerator at a dose of 80 cGy daily, starting 11 days before transplantation, until a total of 10 doses (800 cGy) has been delivered. The irradiation will consist of a supradiaphragmatic mantle field, a subdiaphragmatic field including an inverted Y and splenic ports, encompassing all major lymphoid organs, including the thymus, spleen, and lymph nodes, as used in the treatment of Hodgkin's disease (Kaplan HS, Cancer Research 26:1268-1276, 1966). The Waldeyer ring is not included. ATG (Thymoglobulin®, Genzyme), at a dose of 1.5 mg/kg/d, will be given intravenously on days -11 through -7.
  Conditioning regimen II (TLI 8 Gy + ATG [Thymoglobulin]): TLI 8 Gy + ATG (Thymoglobulin) 7.5 mg/kg
Period: Overall Study
Arm/Group | Flu-TBI | TLI-ATG
Started | 50 (5 patients in Screening failure between inclusion and transplantation) | 47 (5 patients in Screening failure between inclusion and transplantation)
Completed | 49 | 45
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Population: 13/107 included patients (6 in the Flu-TBI and 7 in the TLI-ATG arm) were excluded from analysis because they did not meet the inclusion criteria at the time of the start of the conditioning (disease relapse (5), ineligible for further irradiation (3), donor refusal (2), HLA-mismatched donor (2), and poor PS (1)).
Groups:
- Total: Total of all reporting groups
Arm/Group | Flu-TBI | TLI-ATG | Total
Number analyzed (Participants) | 49 | 45 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 35 | 71
  >=65 years | 13 | 10 | 23
Age, Continuous [Median (Full Range); unit: years] | 60 [38 to 73] | 59 [32 to 71] | 60 [32 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 35 | 29 | 64
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 4 | 2 | 6
  Belgium | 45 | 43 | 88
Donor: HLA-identical sibling/ 10/10 HLA-allele matched URD [Number; unit: participants]
  HLA-identical sibling | 29 | 25 | 54
  10/10 HLA-allele matched URD | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade II-IV Acute GVHD Between the 2 Groups
Description: Percentage of participants with aGVHD according grades:
  Grade I: rash skin < 25 % area; bilirubin: 20-30 mg/ml; diarrhea: 500-1000 ml/day Grade II: rash skin 25-50 % area; bilirubin: 30-60 mg/ml; diarrhea: 10000-1500 ml/day Grade III:rash skin > 50 % area; bilirubin: 60-150 mg/ml; diarrhea: >1500 ml/day Grade IV: erythroderma; bilirubin: > 150 mg/ml; diarrhea: >2000 ml/day
  Grade IV is the worst grade Patients given a second allogeneic HCT were censured for GVHD analyses.
Time Frame: 180 days after HCT
Population: Patients given a second allogeneic HCT were censured for GVHD analyses.
Measure: Number; unit: percentage of participants with aGVHD
Arm/Group | Flu-TBI | TLI-ATG
Number analyzed (Participants) | 48 | 40
percentage of participants with aGVHD | 12.2 | 8.9
Statistical Analysis 1: Comparison: Flu-TBI vs TLI-ATG; Test type: Superiority; p = 0.508, Multivariate Cox models
Statistical Analysis 2: Comparison: Flu-TBI vs TLI-ATG; At day 180; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Flu-TBI vs TLI-ATG; At Day 365; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants With Graft Rejection as Defined by Whole Blood and T Cell Chimerism
Description: graft rejection are reported in outcome measure data table (defined as ≤ 5% donor chimerism in T cells, total white blood cells and/or total bone marrow cells).
Time Frame: 1 year after HCT
Measure: Number; unit: participants
Arm/Group | Flu-TBI | TLI-ATG
Number analyzed (Participants) | 49 | 45
participants | 3 | 4
Statistical Analysis 1: Comparison: Flu-TBI vs TLI-ATG; At day 100; Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Flu-TBI vs TLI-ATG; At Day 40; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Flu-TBI vs TLI-ATG; At Day 180; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percentage of Participants With Chronic GVHD in the 2 Groups
Description: Comparaison of the number of Participants with chronic GVHD in the 2 groups
Time Frame: 2 years after HCT
Population: Patients given a second allogeneic HCT were censured for GVHD analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Flu-TBI | TLI-ATG
Number analyzed (Participants) | 48 | 40
percentage of participants | 40.8 | 18.8
Statistical Analysis 1: Comparison: Flu-TBI vs TLI-ATG; Test type: Superiority; p = 0.0165, Multivariate Cox models
Statistical Analysis 2: Comparison: Flu-TBI vs TLI-ATG; Test type: Superiority; p = 0.010, Mutivariate; Hazard Ratio (HR) = 0.3
Statistical Analysis 3: Comparison: Flu-TBI vs TLI-ATG; Test type: Superiority; p = 0.0495, Multivariate; Hazard Ratio (HR) = 0.5
Statistical Analysis 4: Comparison: Flu-TBI vs TLI-ATG; Test type: Superiority; p = 0.001, Multivariate; Hazard Ratio (HR) = 3.8

4. Secondary Outcome: Incidences of Bacterial, Fungal and Viral Infections in the 2 Groups.
Time Frame: D100 after HCT
Measure: Number; unit: participants
Arm/Group | Flu-TBI | TLI-ATG
Number analyzed (Participants) | 49 | 45
participants
  Bacterial infection | 19 | 25
  Fungal infection | 3 | 7
  CMV reactivation | 15 | 21
Statistical Analysis 1: Comparison: Flu-TBI vs TLI-ATG; 19 of 49 Flu-TBI patients (39%) versus 25 of 45 TLI ATG patients (56%) had a least one episode of bacterial infection the first 100 days after transplantation (P = 0.15); Test type: Superiority; p = 0.15, Fisher Exact
Statistical Analysis 2: Comparison: Flu-TBI vs TLI-ATG; For fungal infections, the figures were 3 of 45 (6%) and 7 of 45 (16%), respectively (P = 0.19); Test type: Superiority; p = 0.19, Fisher Exact
Statistical Analysis 3: Comparison: Flu-TBI vs TLI-ATG; Among CMV-seropositive patients and/or donors, the 100-day cumulative incidence of CMV reactivation was 31% in Flu-TBI patients versus 47% in TLI-ATG patient; Test type: Superiority; p = 0.12, Fisher Exact

5. Secondary Outcome: Percentage of Relapse Rate in the 2 Groups
Time Frame: 1 year after HCT
Measure: Number; unit: percentage of Relapse
Arm/Group | Flu-TBI | TLI-ATG
Number analyzed (Participants) | 49 | 45
percentage of Relapse | 22 | 50
Statistical Analysis 1: Comparison: Flu-TBI vs TLI-ATG; Four-year cumulative incidences of relapse/progression were 22% and 50% in Flu-TBI and TLI-ATG patients, respectively; Test type: Superiority; p = 0.017, Cumulative incidence curves; Multivariate Cox models = 2.3, 95% CI 2-sided [1.1 to 4.7], Standard Deviation 0.02

6. Secondary Outcome: Quality and Timing of Immunologic Reconstitution: Concentration of ATG Levels
Description: Analyses of ATG levels in order to assess the immune system recuperation
Time Frame: Day 0, Day 3 and Day 10
Measure: Median (95% Confidence Interval); unit: mg/L
Arm/Group | TLI-ATG
Number analyzed (Participants) | 15
mg/L
  Median ATG serum levels at day 0 | 4 [3.8 to 4.2]
  Median ATG serum levels at day 3 | 2.2 [2.09 to 2.31]
  Median ATG serum levels at day 10 | 0.95 [0.9025 to 0.9975]
Statistical Analysis 1: Comparison: TLI-ATG; This statistical analysis applies to median ATG serum levels at day 0; Test type: Superiority; Median Difference (Final Values) = 4
Statistical Analysis 2: Comparison: TLI-ATG; This statistical analysis applies to median ATG serum levels at day 3; Test type: Superiority; Mean Difference (Final Values) = 2.2
Statistical Analysis 3: Comparison: TLI-ATG; This statistical analysis applies to median ATG serum levels at day 10; Test type: Superiority; Mean Difference (Final Values) = 0.95

7. Secondary Outcome: Percentage of Non Relapse Mortality in the 2 Groups
Time Frame: 1 year after HCT
Measure: Number; unit: percentage of participants
Arm/Group | Flu-TBI | TLI-ATG
Number analyzed (Participants) | 49 | 45
percentage of participants | 24 | 13
Statistical Analysis 1: Comparison: Flu-TBI vs TLI-ATG; Test type: Superiority; p = 0.5, Cumulative incidence curve

8. Secondary Outcome: Percentage of 4-year Progression Free Survival in the 2 Groups
Time Frame: 4 year after HCT
Measure: Number; unit: percentage of participants
Arm/Group | Flu-TBI | TLI-ATG
Number analyzed (Participants) | 49 | 45
percentage of participants | 54 | 37
Statistical Analysis 1: Comparison: Flu-TBI vs TLI-ATG; Test type: Superiority; p = 0.14, Kaplan-Meier method; multivariate analyses = 2, 95% CI 2-sided [1 to 4.1], Standard Deviation 0.07

9. Secondary Outcome: Percentage of 5-year Progression Free Survival in the 2 Groups
Time Frame: 5 year after HCT
Measure: Number; unit: percentage of participants
Arm/Group | Flu-TBI | TLI-ATG
Number analyzed (Participants) | 49 | 45
percentage of participants | 50 | 37

10. Secondary Outcome: Percentage of 4-year Overall Survival in the 2 Groups
Time Frame: 4 year after HCT
Measure: Number; unit: percentage of participants
Arm/Group | Flu-TBI | TLI-ATG
Number analyzed (Participants) | 49 | 45
percentage of participants | 53 | 54
Statistical Analysis 1: Comparison: Flu-TBI vs TLI-ATG; Test type: Superiority; p = 0.9, Kaplan-Meier method; multivariate analyses = 1.2, 95% CI 2-sided [1 to 1.4], Standard Deviation 0.02

11. Secondary Outcome: Percentage of 5-year Overall Survival in the 2 Groups
Time Frame: 5 year after HCT
Measure: Number; unit: percentage of participants
Arm/Group | Flu-TBI | TLI-ATG
Number analyzed (Participants) | 49 | 45
percentage of participants | 53 | 55
Statistical Analysis 1: Comparison: Flu-TBI vs TLI-ATG; Test type: Superiority; p = 0.96, Kaplan-Meier method; multivariate analyses = 1.2, 95% CI 2-sided [1 to 1.4], Standard Deviation 0.02

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Flu-TBI | TLI-ATG
All-Cause Mortality (participants affected / at risk) | 22/49 | 19/45
Serious Adverse Events (participants affected / at risk) | 41/49 | 41/45
Other Adverse Events (participants affected / at risk) | 15/49 | 21/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flu-TBI (N=49) | TLI-ATG (N=45)
acute Graft versus Host Disease (Immune system disorders) | 5 | 5
chronic Graft versus Host Disease (Immune system disorders) | 20 | 13
Graft failure (Blood and lymphatic system disorders) | 3 | 4
Relapse/progression (Blood and lymphatic system disorders) | 12 | 22
Acute respiratory distress syndrom (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — ARDS
Lung (Infections and infestations) | 7 | 2
Septic shock (Infections and infestations) | 5 | 5
Second maligancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Viral infection (Infections and infestations) | 6 | 4
Fever unknown origin (General disorders) | 3 | 5 — FUO
Multiple organ failure (General disorders) | 0 | 1 — MOF
surgical procedure (Surgical and medical procedures) | 2 | 3 — planed surgery, biopsy, endoscopy
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Catheter (Infections and infestations) | 2 | 0
Urinary tract (Infections and infestations) | 2 | 0
GI complains (Gastrointestinal disorders) | 4 | 3 — anorexia, pain, gastroenteritis
Neurologic troubles (Nervous system disorders) | 4 | 1 — pain, depression, sleeping trouble
Epilepsy (Nervous system disorders) | 1 | 0
Hemolytic anemia (Blood and lymphatic system disorders) | 0 | 1
Alveolar Hemorrhage (Blood and lymphatic system disorders) | 1 | 1
Hematuria (Blood and lymphatic system disorders) | 0 | 1
Acute renal failure (Renal and urinary disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flu-TBI (N=49) | TLI-ATG (N=45)
CMV reactivation (Infections and infestations) | 15 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No